CLINICAL TRIAL: NCT03324789
Title: Comparative Study Between Single Implant Retained Partial Over-denture and Conventional Partial Denture in Mandibular Long Span Kennedy Class IV ( Randomized Clinical Trial )
Brief Title: Comparison Between Single Implant Retained Partial Over-denture and Conventional Partial Denture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Radwa Ahmed Abdel Wanis, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9999
Record Dates: First submitted 2017-10-02; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Bone Loss in Jaw
Keywords: Single implant; Anterior edentulism; partial denture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding will only be done for the outcome assessor for patient satisfaction and the statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Implant Partial Over-denture (Experimental): The design will be as follows; two rests on principle abutments and lingual plate major connector, single implant in the symphyseal region.
  Interventions: Other: Single Implant Partial Over-denture
- Conventional Partial Denture (Active Comparator): patients will receive conventional partial denture with double Aker clasp on mandibular second premolar and first molar, with no indirect retention and lingual plate as major connector .
  Interventions: Other: Conventional Partial Denture

INTERVENTIONS:
Other: Single Implant Partial Over-denture — Single Implant Retained Partial Over-denture will be as follows; two rests on principle abutments and lingual plate major connector, single implant in the symphyseal region.
  Arms: Single Implant Partial Over-denture
Other: Conventional Partial Denture — patients will receive conventional partial denture with double Aker clasp on mandibular second premolar and first molar, with no indirect retention and lingual plate as major connector .
  Arms: Conventional Partial Denture

SUMMARY:
In this study we are going to evaluate patient satisfaction as well as the amount of bone loss on using single implant retained partial over-denture versus conventional partial denture for treatment of mandibular Kennedy class IV cases

DETAILED DESCRIPTION:
All the procedures will be made in the outpatient clinic of the removable prosthodontics department, faculty of oral medicine, Cairo University except the CBCT will be performed in the Oral radiology department, faculty of oral medicine, Cairo University.

The selected patients will be informed of the nature of the research work and informed consent will be signed by each one of them. Only motivated patients who showed co-operation will participate in the study. Patients will be randomly divided into 2 groups.

Clinical examination and investigations will be carried out for the eligible patients including TMJ examination and intraoral examination for oral mucosa. Diagnostic charts will be prepared with full medical and dental history as well as radiographic records. The upper and lower study casts were mounted on a semi-adjustable articulator to evaluate the interarch space and the occlusal plane.

Abutment teeth will be evaluated regarding mobility, caries, existing restoration, over eruption, and malalignment. Pocket depth around the abutment teeth will be measured buccally, lingually, and proximally. Radiographic evaluation of all abutment teeth will be carried out to assess the amount of bone support, crestal bone height, continuity of lamina dura, periapical pathosis, crown/root ratio, and root form. Panoramic radiograph also to evaluate the bone quality and quantity in the lower anterior region.

All the patients will be motivated for meticulous oral hygiene.

In (Group I) The design of the finished partial overdenture will be as follows; two rests on principle abutments and lingual plate major connector. The trial of the metallic framework will be carried out for proper seat and fit.

Patients will receive anterior single implant in the mandibular sympheseal region.

The locator attachment will be inserted into the implant fixture, leaving the attachment base protruding at least 2 mm above the tissue surface. The partial overdenture will be filled with resin, and the patient will be guided to occlude in centric occlusion. The partial overdenture will be removed after the resin curing and adjusted accordingly to assure a comfortable fit.

In (Group2) The design of the finished removable partial denture will be as follows; double Aker clasp on mandibular second premolar and first molar, with no indirect retention and lingual plate as major connector .

ELIGIBILITY:
Inclusion Criteria:

* Mandibular long span Kennedy class IV patients
* Patients with full set of opposing dentition
* Patients having enough implant bone height
* No apparent bony mal-relation.
* No intraoral soft or hard tissue pathosis
* No uncontrolled systemic diseases such as hypertension, diabetes and immunodeficiency.

Exclusion Criteria:

* Drug or alcohol abuse
* A health condition precluding surgery
* Physical reasons that could affect follow-up
* Psychiatric problems
* Disorders to the implant area related to a history of radiation therapy to the head and neck, neoplasia, or bone augmentation to the implant site.
* Heavy smokers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | six months
  will be measured using Visual Analogue Scale (VAS) , represented by a horizontal line 100 mm in length where the patient marks on the line the point that best represents their current state where the severity increases from the left to the right side of the line & it's degree is marked according to their answers to a questionnaire of five questions prepared on how well satisfied they are with the new treatment they are receiving

SECONDARY OUTCOMES:
Bone loss | Nine months
  Bone height will be measured in millimeters using DIGORA machine Digital subtraction radiography will be used where Dental images will be obtained before & after implant placement using the paralleling technique, Bone height will be measured at denture delivery, 4, 9 months respectively after denture insertions

CONTACTS AND LOCATIONS:
Overall Officials: Radwa Sheta, Principal Investigator — Faculty of dentistry-Cairo Uni
Locations (1):
- Faculty of dentistry-Cairo Uni, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided